CLINICAL TRIAL: NCT00975338
Title: The LETS Study: A Longitudinal Evaluation of Transition Services
Acronym: LETS
Status: Completed | Type: Observational
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Ontario Neurotrauma Foundation (Other)
Responsible Party: Principal Investigator, Shauna Kingsnorth, Clinical Study Investigator, Bloorview Research Institute, The Hospital for Sick Children
Other Study IDs: 2008-ABI-LSMODEL-706
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Cerebral Palsy; Brain Injuries; Spinal Dysraphism
Keywords: health care transition, young adults, rehabilitation
MeSH Terms: conditions — Cerebral Palsy; Brain Injuries; Spinal Dysraphism | interventions — Longevity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Prospective LIFEspan: LIFEspan youths with Cerebral Palsy or Acquired Brain Injury
  Interventions: Other: LIFEspan
- Prospective Non-LIFEspan: LIFEspan youths with Spina Bifida
  Interventions: Other: Non-LIFEspan
- Retrospective Non-LIFEspan: Non-LIFEspan youths with Cerebral Palsy or Acquired Brain Injury
  Interventions: Other: Non-LIFEspan
- LIFEspan Staff: All staff affiliated with the LIFEspan model of linked transition care
  Interventions: Other: LIFEspan
- Caregivers: Parents of participating youths
  Interventions: Other: LIFEspan

INTERVENTIONS:
Other: LIFEspan — Rehabilitation services provided by an inter-disciplinary team of health professionals addressing the transfer of care to adult services and emerging needs related to transition to adulthood. LIFEspan staff are cross-appointed to both a pediatric and an adult hospital through a formally linked model of care.
  Other Names: LIFEspan model of linked transition care
  Groups: Caregivers; LIFEspan Staff; Prospective LIFEspan
Other: Non-LIFEspan — Standard of care in the absence of a formal partnership between a pediatric and an adult hospital.
  Groups: Prospective Non-LIFEspan; Retrospective Non-LIFEspan

SUMMARY:
This project will describe and evaluate the impact of a unique partnership model designed to coordinate transfer of care by formally linking pediatric and adult heath care services. The experiences of young people receiving this model of care will be compared and contrasted against the experiences of young people receiving the current standard of care. Young people with a diagnosis of Cerebral Palsy (CP), Acquired Brain Injury in childhood (ABIc), and Spina Bifida (SB) will be followed during the transition period. Preparation for transition, health care, and transfer of care service delivery will be detailed in a process evaluation. An outcome evaluation will measure the ability of the two models of service to enable youth to maintain continuity within the health care system after transitioning from pediatric to adult care. Secondary outcomes, including how health, well-being, social participation, transition readiness, and health care utilization are affected will also be explored.

DETAILED DESCRIPTION:
Due to advances in medical treatment, most children with disabilities such as cerebral palsy or acquired brain injury can expect to live normal lifespans. As children, these individuals are cared for by expert healthcare providers working in coordinated teams in specialized pediatric settings. As these children reach adulthood, the availability of services and expertise drops dramatically because the adult health care system has not evolved to meet their specialized needs. In addition, transitioning from pediatric to adult services is often very difficult and stressful. Young people and their families must leave familiar healthcare settings and providers, and secure care in unfamiliar adult health care environments.

This proposed project will describe and evaluate the impact of a unique partnership model designed to coordinate transfer of care by formally linking pediatric and adult health care services. The LIFEspan model aims to (a) prepare youth and their families to adapt to adult healthcare provision, (b) provide a coordinated transfer process from pediatric to adult providers, and (c) establish sustainable access and appropriate adult care. The project will detail the specific service delivery that occurs with respect to preparation for transition and transfer of care in a process evaluation. An outcome evaluation will measure the effectiveness of the model in terms of its abilities to enable youth to maintain continuity within the health care system after transitioning from pediatric to adult care. Secondary outcomes, including how health, well-being, social participation, transition readiness, and health care utilization are affected by the LIFEspan model, will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Prospective groups: 16th Birthday between September 2008 - August 2009, diagnosis of cerebral palsy or acquired brain injury, spina bifida
* Retrospective group: 16th Birthday between September 2002 - August 2003, diagnosis of cerebral palsy or acquired brain injury

Exclusion Criteria:

* N/A

Ages: 16 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Youth and young adult clients or recent graduates of Bloorview Kids Rehab who have either participated in LIFEspan transition services or have transitioned to adult healthcare without LIFEspan participation
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2016-07-12 (Actual)

PRIMARY OUTCOMES:
maintenance of continuous care | September 2009 - September 2013

SECONDARY OUTCOMES:
patterns of health care utilization, health, well-being, social participation and transition readiness | September 2009 - September 2013

CONTACTS AND LOCATIONS:
Overall Officials: Colin Macarthur, PhD, Principal Investigator — The Hospital for Sick Children; Mark Bayley, MD, Principal Investigator — Toronto Rehab Institute
Locations (2):
- Canada (2):
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario
  - Toronto Rehabilitation Institute, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsybina I, Kingsnorth S, Maxwell J, Bayley M, Lindsay S, McKeever P, Colantonio A, Hamdani Y, Healy H, Macarthur C. Longitudinal Evaluation of Transition Services ("LETS Study"): protocol for outcome evaluation. BMC Pediatr. 2012 May 15;12:51. doi: 10.1186/1471-2431-12-51. PMID 22587415
- [Result] Kingsnorth, S., Lindsay, S., Maxwell, J., Tsybina, I., Seo, H., Macarthur, C., & Bayley, C. (2011). Implementing the LIFEspan model of transition care for youth with childhood onset disabilities. International Journal of Adolescent & Child Health, 3(4), 547-560.https://www.novapublishers.com/catalog/product _info.php?products_id=23001
- [Result] Hamdani Y, Proulx M, Kingsnorth S, Lindsay S, Maxwell J, Colantonio A, Macarthur C, Bayley M. The LIFEspan model of transitional rehabilitative care for youth with disabilities: healthcare professionals' perspectives on service delivery. J Pediatr Rehabil Med. 2014;7(1):79-91. doi: 10.3233/PRM-140271. PMID 24919941
- [Result] Lindsay S, Proulx M, Maxwell J, Hamdani Y, Bayley M, Macarthur C, Colantonio A. Gender and Transition From Pediatric to Adult Health Care Among Youth With Acquired Brain Injury: Experiences in a Transition Model. Arch Phys Med Rehabil. 2016 Feb;97(2 Suppl):S33-9. doi: 10.1016/j.apmr.2014.04.032. Epub 2015 Feb 4. PMID 25660004
- [Result] Kingsnorth S, Lindsay S, Maxwell J, Hamdani Y, Colantonio A, Zhu J, Bayley MT, Macarthur C. Bridging Pediatric and Adult Rehabilitation Services for Young Adults With Childhood-Onset Disabilities: Evaluation of the LIFEspan Model of Transitional Care. Front Pediatr. 2021 Sep 17;9:728640. doi: 10.3389/fped.2021.728640. eCollection 2021. PMID 34631624
- [Result] Kingsnorth S, Hamdani Y, Cheng C, Lindsay S, Maxwell J, Colantonio A, Bayley M, Macarthur C. Health status and health care utilization profiles of adolescents with disabilities. Health Care Transit. 2023 Jun 21;1:100004. doi: 10.1016/j.hctj.2023.100004. eCollection 2023. PMID 39713020